CLINICAL TRIAL: NCT00414804
Title: Spinal Cord Stimulation (SCS) Versus Nerve Blocks and Physical Therapy for Complex Regional Pain Syndrome
Brief Title: Spinal Cord Stimulation Versus Nerve Blocks and Physical Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decided to withdraw participation in the study
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCS0805
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Complex Regional Pain Syndrome; Chronic Pain; Pain
Keywords: Pain; Neurostimulation
MeSH Terms: conditions — Complex Regional Pain Syndromes; Chronic Pain; Pain | interventions — Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal Cord Stimulation (SCS) Group (Active Comparator): Spinal Cord Stimulation (SCS) Treatment Group
  Interventions: Device: Precision SCS
- Nerve Blocks and PT (Active Comparator)
  Interventions: Procedure: Nerve Blocks and PT

INTERVENTIONS:
Device: Precision SCS — Precision Spinal Cord Stimulation (SCS) Therapy
  Arms: Spinal Cord Stimulation (SCS) Group
Procedure: Nerve Blocks and PT — Pain therapy utilizing Nerve Blocks with Physical Therapy
  Arms: Nerve Blocks and PT

SUMMARY:
The primary objective of this study is to compare the efficacy of SCS using the Precision implantable neurostimulation device and conventional medical treatment (nerve blocks + physical therapy) in subjects with recently-diagnosed Complex Regional Pain Syndrome (CRPS) after some more conservative treatments have failed. There are significant numbers of patients with CRPS in whom conventional treatment is ineffective and SCS is used only as a last resort. If SCS is effective earlier in the treatment continuum, it would provide a much needed treatment alternative and increase awareness of the utility of SCS for this indication. It is also possible that early intervention with SCS may limit disease progression.

DETAILED DESCRIPTION:
Standard medical treatment for moderate/severe chronic pain of Complex Regional Pain Syndrome (CRPS) is usually inadequate. Sympathetic nerve blocks with local anesthetics are commonly employed and in some cases can be an effective option. Nerve blocks are not consistently effective, however, and their utility is further compromised by a short duration of relief.

CRPS is among the pain etiologies that can be managed via Spinal Cord Stimulation (SCS); this option can be quite effective at providing long-term pain relief for the management of CRPS. Importantly, SCS is not usually attempted until other treatment options, including nerve blocks and ablative procedures, have failed to produce adequate pain relief. No studies have been performed to date comparing SCS to a series of nerve block injections plus physical therapy. In this context, it may be prudent to consider SCS earlier in the treatment continuum. Instead of obliging a CRPS patient to cycle through numerous rounds of injections, optimal clinical pain management may be attained through early implantation of an SCS system. This prospective clinical study will compare the relative efficacy of SCS with that of repeated nerve blocks and physical therapy in a group of subjects with moderate-to-severe CRPS pain.

Patients who have never had invasive treatments for CRPS pain will be randomized to either a series of sympathetic blocks plus physical therapy or SCS. Changes in pain, disability, and quality of life outcomes will be assessed at follow up visits as well as incidence and outcomes of subjects electing to cross over to the alternate treatment option. This study will generate insight into the best pain management strategies for CRPS.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with chronic CRPS with intractable neuropathic pain of moderate to severe intensity within the last 3-6 months.
* Have failed initial treatment for CRPS, such as physical therapy alone, oral medications, and/or steroids.
* Be 18 years of age or older.
* Be an appropriate candidate for the surgical procedures required for SCS.
* Be willing and able to comply with all study related procedures and visits.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have had any unsuccessful back or spine surgery that currently causes pain.
* Have had any treatment for CRPS other than physical therapy, oral medications, or steroids.
* Have any evidence of neurologic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
The primary endpoint is reduction in baseline levels of pain; | 12-weeks post SCS treatment compared to Nerve Blocks+PT

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Simopoulos, MD, Principal Investigator — Beth Israel Deaconess Medical Center